CLINICAL TRIAL: NCT01598467
Title: Prospective Interventional Study on Robotic Sacrocolpopexy: a European Multicentric Cohort (PARSEC)
Brief Title: Prospective Assessment of Robotic Sacrocolpopexy: a European Multicentric Cohort (PARSEC)
Acronym: PARSEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Femke van Zanten (Other)
Responsible Party: Sponsor-Investigator, Femke van Zanten, Study Coordinator, urologist, urogynaecology fellow, Cork University Hospital
Organization: Cork University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PARSEC-1
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; POP; sacrocolpopexy; sacrohysteropexy; promontofixation; colpopexy; robotic surgery; surgical complications; mesh; prolapse repair
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Women with pelvic organ prolapse (Other): Women with pelvic organ prolapse (simplified POP-Q > stage 1)
  Interventions: Procedure: Robotic assisted sacrocolpopexy (RASC)

INTERVENTIONS:
Procedure: Robotic assisted sacrocolpopexy (RASC) — Robotic assisted sacrocolpopexy (RASC) will be performed with the Da Vinci Surgical robot (Intuitive Surgical). THe mesh used will be a Type I (Amid classification), polypropylene mesh
  Other Names: sacrocolpopexy, colpopexy, promontofixation, hysteropexy, colposacrohysteropexy, sacropexy

SUMMARY:
The purpose of this study is to prospectively assess the outcomes of robotic sacrocolpopexy for repair of pelvic organ prolapse in high volume european centers.

DETAILED DESCRIPTION:
To prospectively assess the outcomes of robotic sacrocolpopexy for repair of pelvic organ prolapse in high volume european centers.

Primary outcome: anatomical cure rate (using simplified POP-Q staging system)

Secondary outcomes:

complication assessment (Clavien-Dindo), functional results, intraoperative variables, impact of surgery on quality of life (PFIQ-7, PISQ-12)

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic vaginal vault prolapse with simplified pelvic organ prolapse quantification (POP-Q) stage 2 or greater

Exclusion Criteria:

* Poor health status with inability to undergo general anaesthesia
* Age < 18 years
* ≥ 3 previous laparotomic surgeries
* Planned pregnancy
* Other: known pelvic malignancies, previous pelvic radiotherapy, congenital anomalies of genitourinary tract, autoimmune diseases with connective tissue involvement (Lupus, Sjogren Sdr, sclerodermia, etc.), current UTI's, use of steroids, anticoagulants, interstitial cystitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
anatomical cure after robotic assisted sacrocolpopexy (or absence of recurrent prolapse) | 6 months
  anatomical cure (defined as any simplified POP-Q point <2) will be assessed at regular intervals(see time frame). If any postoperative POP-Q point will be ≥2, this will be recorded as a recurrent prolapse.

SECONDARY OUTCOMES:
intra- peri- and postoperative complications | intraoperative to 6 weeks after surgery
  complications occurring during surgery are defined as "intraoperative complication", within 3 weeks from surgery will be defined as "perioperative complication". Complications occurring after this timeframe will be regarded as "late complications", if related to surgery (e.g. mesh erosion)
quality of life | 6 weeks, 6 months, 1 year (yearly thereafter, if feasible)
  impact of prolapse repair on quality of life will be assessed via specific validated questionnaires (PFIQ-7, PISQ-12)
postoperative pain | on postoperative day 1
  pain will be assessed on a visual analogue scale (range 0 to 10= 0 no pain, 10 unbearable pain)
intraoperative variables | intraoperative
  intraoperative variables are recorded, such as: blood loss, duration of surgery (divided in robotic setup time, console time and surgery completion time). Concomitant procedures, such as adhesiolysis will also be recorded
impact of uterus management | 6 weeks, 6 months, 1 year (yearly thereafter, if feasible)
  logistic regression analysis will be performed to evaluate if different surgical approaches in presence, -or absence, of the uterus (e.g. supracervical hysterectomy, uterus sparing surgery), have an effect on primary and secondary outcomes
anatomical cure after robotic assisted sacrocolpopexy (or absence of recurrent prolapse) | 6 weeks
  anatomical cure (defined as any simplified POP-Q point <2) will be assessed at regular intervals(see time frame). If any postoperative POP-Q point will be ≥2, this will be recorded as a recurrent prolapse.
anatomical cure after robotic assisted sacrocolpopexy (or absence of recurrent prolapse) | 1 year, yearly thereafter (if feasible)
  anatomical cure (defined as any simplified POP-Q point <2) will be assessed at regular intervals(see time frame). If any postoperative POP-Q point will be ≥2, this will be recorded as a recurrent prolapse.

CONTACTS AND LOCATIONS:
Overall Officials: Barry O'Reilly, Principal Investigator — Cork University Hospital; Steven E Schraffordt Koops, Study Chair — Department of Gynecology and Obstetrics, Meander Medical Center, Amersfoort, The Netherlands; Lorenzo Dutto, Study Chair — Cork University Hospital
Locations (1):
- Cork University Maternity Hospital, Cork, Ireland

REFERENCES:
- [Derived] van Zanten F, Schraffordt Koops SE, O'Sullivan OE, Lenters E, Broeders I, O'Reilly BA. Robot-assisted surgery for the management of apical prolapse: a bi-centre prospective cohort study. BJOG. 2019 Jul;126(8):1065-1073. doi: 10.1111/1471-0528.15696. Epub 2019 May 2. PMID 30924606